CLINICAL TRIAL: NCT04654806
Title: Assessment of Left Ventricular Diastolic Function in Patients With Atrial Fibrillation
Acronym: DIAAF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2020-1105
Record Dates: First submitted 2020-11-26; First posted 2020-12-04 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a single-center, prospective cohort study to investigate non-invasive method to assess left ventricular diastolic function using echocardiography. Patients with AF who are referred radiofrequency catheter ablation (RFA) will be included prospectively. Transthoracic echocardiography will be performed during, immediately before RFA and with no cardiovascular medication taken between the exams so that the loading conditions during catheterization and echocardiography are as similar as possible. We will validate previously proposed echocardiographic parameters and creat an algorithm to identify the relationship between echocardiographic parameters of diastolic function and invasively measured LA pressure in patients with atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 19 year-old
* Patients who scheduled to perform radiofrequency catheter ablation for atrial fibrillation
* Patients who had paroxysmal, persistent, or chronic AF
* Patients provided with the written, informed consent to participate in this study

Exclusion Criteria:

* Patients with prosthetic valve
* Life expectancy < 12 months
* Subject who the investigator deems inappropriate to participate in this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who scheduled to perform radiofrequency catheter ablation for atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-11-25 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Association between mean left atrial pressure and echocardiographic parameters | up to 12 weeks after collecting all data
  Correlation between echocardiographic parameters or algorithm to estimate invasively measured left atrial pressure.
  Echocardiographic parameters: E/A ratio, E velocity, e' velocity, E/e', IVRT. LV strain, RV strain,, LA strain, Vp, E/Vp, LA volume index, TV V max, and Peak acceleration rate of mitral E velocity

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Won Ha, Principal Investigator — Severance Hospital
Locations (1):
- Division of Cardiology, Severance Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No